CLINICAL TRIAL: NCT01585935
Title: Preventing Cholestasis in Premature Infants Using SMOFLipid®
Brief Title: Preventing Cholestasis Using SMOFLipid®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoc.Prof.MD., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MUV-Neo2; 2011-005456-33 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-26 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Cholestasis; Psychomotor Disorders, Developmental
Keywords: Infant, Extremely Low Birth Weight; Parenteral Nutrition; Fish Oils; Cholestasis; Psychomotor Disorders, Developmental
MeSH Terms: conditions — Cholestasis; Psychomotor Disorders; Hyperphagia | interventions — SMOFlipid; In Situ Hybridization, Fluorescence; Olive Oil; soybean oil, phospholipid emulsion; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoflipid (Experimental): SMOFLIPID will be used for parenteral lipid supply
  Interventions: Drug: SMOFLIPID
- Intralipid (Active Comparator): INTRALIPID will be used for parenteral lipid supply
  Interventions: Drug: INTRALIPID

INTERVENTIONS:
Drug: SMOFLIPID — target dose: 3g/kg/d
  Other Names: SMOFLIPID (mixture of soy, fish, MCT and olive oil)
  Arms: Smoflipid
Drug: INTRALIPID — target dose: 3g/kg/d
  Other Names: INTRALIPID (soy bean oil)
  Arms: Intralipid

SUMMARY:
Preterm infants of extreme low birth weight (ELBW, < 1000 gram birth weight) cannot immediately be nourished with mother´s or formula milk and are typically dependent on parenteral nutrition (PN) for a prolonged period of time. This puts them at risk for liver complications of PN, namely parenteral nutrition associated cholestasis (PNAC).

Intravenous lipid emulsions (ILE) based on soy bean oil are standard of care for provision of energy and essential fatty acids in preterm infants. However, they might be implicated in the pathogenesis of PNAC.

ILEs based on pure fish oil are proposed for therapy of PNAC. Recently a lipid emulsion containing 15 % fish oil together with soy bean, olive and MCT oil has become available in Europe (SMOFLIPID®). Such a balanced lipid emulsion might be more favourable than the standard soy bean oil emulsion (Intralipid®) concerning the development of PNAC. Furthermore ILEs containing fish oil might exert a positive effect on neurodevelopment. However, there are no data so far.

The study aims to evaluate the fish oil containing ILE "SMOFlipid®" for its protective effect against PNAC in ELBW infants compared to standard treatment with the soy bean based ILE "Intralipid®". Furthermore neurodevelopment at 12 and 24 months of corrected gestational age will be investigated.

DETAILED DESCRIPTION:
BACKGROUND: Extreme low birth weight infants (ELBW, < 1000 gram birth weight) are typically dependent on parenteral nutrition (PN) for a prolonged period of time. This puts them at risk for development of liver complications of PN, namely parenteral nutrition associated cholestasis (PNAC).

Intravenous lipid emulsion (ILE) based on soy bean oil are standard of care in preterm infants, but might be implicated in the pathogenesis of PNAC. Fish oil is rich in omega-3 long chain polyunsaturated fatty acids (LC-PUFA) that particularly accumulate in liver and brain of the fetus during the last trimester of pregnancy. In pediatric patients, ILEs based on pure fish oil are proposed as a rescue therapy of PNAC.

Recently a mixed lipid emulsion containing 15 % fish oil together with soy bean , olive and MCT oil has become available for PN in Europe. Such a balanced lipid emulsion might be more favourable than the standard soy bean oil emulsion (Intralipid®) concerning the development of PNAC. Furthermore ILEs containing fish oil might exert a positive effect on neurodevelopment. However there are no data so far.

AIM: To evaluate a fish oil containing ILE (SMOFlipid®) for its prophylactic effect on PNAC in ELBW infants compared to a soy bean based ILE (Intralipid®).

STUDY DESIGN: Double blind prospective randomized trial.

* Primary Outcome: PNAC defined as two conjugated bilirubin > 1.5 mg/dl measurements on two consecutive occasions.
* Secondary Outcome: The most important secondary outcome is neurodevelopment at 12 and 24 months of corrected age.
* Exploratory Outcomes: Brain maturation measured by amplitude integrated EEG (aEEG) and flashed visual evoked potentials as available from clinical routine examinations

HYPOTHESIS: The use of a mixed lipid emulsion containing fish oil (SMOFLIPID®) will reduce the incidence of PNAC compared to a standard soy bean oil based lipid emulsion.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≤ 1000 Gram
* Admission to the neonatal ward in the first 24 hours of life
* Informed consent and randomization in the first 5 days of life

Exclusion Criteria:

* Triplets or higher
* Conjugated bilirubin > 1.5 mg/dl before inclusion to the study
* Conditions associated with cholestasis independent of parenteral nutrition, i.e. inborn errors of metabolism, viral infections (cytomegaly virus, HIV, Hep B, Hep C), immune mediated hemolytic disease (Rhesus incompatibility), cystic fibrosis and any other primary cholestatic disease
* Congenital neurological malformations for secondary outcome

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of parenteral nutrition associated cholestasis (PNAC) | Participants will be followed for the duration of hospital stay (expected average 14 weeks)
  PNAC definition: Two consecutive conjugated bilirubin measurements > 1.5 mg/dl

SECONDARY OUTCOMES:
Bailey Scales of Infant Development III | At 12 and 24 months corrected gestational age
  Cognitive, Motor and Language Development

OTHER OUTCOMES:
Brain maturational scores assessed by amplitude integrated EEG (aEEG) | Participants will be followed for the duration of hospital stay (expected average 14 weeks)
  aEEG measurements of study infants performed as a part of clinical routine (as specified in the trial study protocol v 1.0-1.3)
Visual Evoked Potentials (VEP) | Participants will be followed for the duration of hospital stay (expected average 14 weeks)
  VEP measurements of study infants performed as a part of clinical routine (as specified in the trial study protocol v 1.0-1.3)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Repa, MD, Study Director — Medical University Vienna; Nadja Haiden, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
After publication of the trial, we currently plan to share IPD upon personal request.
Supporting Information: Study Protocol
Time Frame: After publication for 10 years.
Access Criteria: We are planning to publish the protocols together with the statistical analysis plan as supplemental information. This however depends on the respective journal. Otherwise please request the study protocol together with the statistical analysis plan from the study director andreas.repa@meduniwien.ac.at

REFERENCES:
- [Derived] Thanhaeuser M, Steyrl D, Fuiko R, Brandstaetter S, Binder C, Thajer A, Huber-Dangl M, Haiden N, Berger A, Repa A. A secondary Outcome Analysis of a Randomized Trial Using a Mixed Lipid Emulsion Containing Fish Oil in Infants with Extremely Low Birth Weight: Cognitive and Behavioral Outcome at Preschool Age. J Pediatr. 2023 Mar;254:68-74.e3. doi: 10.1016/j.jpeds.2022.10.014. Epub 2022 Oct 17. PMID 36257349
- [Derived] Thanhaeuser M, Fuiko R, Oberleitner-Leeb C, Brandstaetter S, Binder C, Thajer A, Huber-Dangl M, Haiden N, Pablik E, Berger A, Repa A. A Randomized Trial of Parenteral Nutrition Using a Mixed Lipid Emulsion Containing Fish Oil in Infants of Extremely Low Birth Weight: Neurodevelopmental Outcome at 12 and 24 Months Corrected Age, A Secondary Outcome Analysis. J Pediatr. 2020 Nov;226:142-148.e5. doi: 10.1016/j.jpeds.2020.06.056. Epub 2020 Jun 23. PMID 32590001
- [Derived] Binder C, Giordano V, Thanhaeuser M, Kreissl A, Huber-Dangl M, Longford N, Haiden N, Berger A, Repa A, Klebermass-Schrehof K. A Mixed Lipid Emulsion Containing Fish Oil and Its Effect on Electrophysiological Brain Maturation in Infants of Extremely Low Birth Weight: A Secondary Analysis of a Randomized Clinical Trial. J Pediatr. 2019 Aug;211:46-53.e2. doi: 10.1016/j.jpeds.2019.03.039. Epub 2019 Apr 25. PMID 31030946
- [Derived] Repa A, Binder C, Thanhaeuser M, Kreissl A, Pablik E, Huber-Dangl M, Berger A, Haiden N. A Mixed Lipid Emulsion for Prevention of Parenteral Nutrition Associated Cholestasis in Extremely Low Birth Weight Infants: A Randomized Clinical Trial. J Pediatr. 2018 Mar;194:87-93.e1. doi: 10.1016/j.jpeds.2017.11.012. Epub 2017 Dec 18. PMID 29269199
- See also: Homepage of the Austrian Science Fund (FWF) — http://www.fwf.ac.at/en/about-the-fwf/corporate-policy/
- See also: Vienna General Hospital, Medical University of Vienna — http://www.meduniwien.ac.at/homepage/service/vienna-general-hospital-akh/en/

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: v 1.0 (2011-11-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT01585935/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: v 1.1 (2012-03-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT01585935/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: v 1.2 (2012-09-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT01585935/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: v 1.3 (2013-08-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT01585935/Prot_SAP_003.pdf